CLINICAL TRIAL: NCT05777317
Title: PDN-SENSORY: A Multi-Center Randomized Controlled Trial to Evaluate Pain and Neurological Function With 10 kHz SCS in Treatment of Painful Diabetic Neuropathy
Brief Title: Pain and Neurological Function Improvements With 10 kHz Spinal Cord Stimulation Treatment of Painful Diabetic Neuropathy
Acronym: PDN-SENSORY
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nevro Corp (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CA2022-2 US PDN-Sensory RCT
Record Dates: First submitted 2023-03-08; First posted 2023-03-21 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Painful Diabetic Neuropathy
Keywords: Diabetic Neuropathy; Spinal Cord Stimulation
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Carubicin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Neurological exam assessors are blinded to treatment assignment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- 10 kHz SCS plus CMM (Experimental): Treatment with high frequency, 10 kHz spinal cord stimulation (SCS) in addition to conventional medical management (CMM)
  Interventions: Device: 10 kHz SCS
- CMM alone (Active Comparator): Treatment with conventional medical management (CMM) alone
  Interventions: Other: CMM alone

INTERVENTIONS:
Device: 10 kHz SCS — Spinal cord stimulation programmed to a frequency of 10 kHz
  Other Names: Nevro HFX therapy programmed to a frequency of 10 kHz or high frequency, 10 kHz SCS
  Arms: 10 kHz SCS plus CMM
Other: CMM alone — Conventional medical management alone
  Arms: CMM alone

SUMMARY:
The purpose of this post-market study is to evaluate changes in pain and neurological function with high frequency, 10 kHz spinal cord stimulation (SCS) therapy in patients with chronic, intractable lower limb pain associated with diabetic peripheral neuropathy, a condition known as painful diabetic neuropathy (PDN). This is a multi-center, prospective, randomized controlled study to evaluate improvement in pain and neurological function in PDN patients, with neurological function assessed via objective measures. Patients will be randomized to conventional medical management (CMM) or 10 kHz SCS plus CMM.

ELIGIBILITY:
Inclusion Criteria:

* Has been clinically diagnosed with diabetes, according to the American Diabetes Association guidelines, as well as painful diabetic neuropathy (PDN) of the lower limbs.
* Has pain intensity (over the last 7 days) of ≥5 out of 10 cm on the Visual Analog Scale (VAS) in the lower limbs at both the Enrollment and Baseline Visits.
* Has PDN symptoms that have been present ≥12 months.
* Is currently taking or has tried in the past a gabapentinoid and at least one other class of analgesic with insufficient pain relief or intolerable side effects.
* Has been on a stable analgesic regimen, as determined by the Investigator, for at least 30 days prior to assessing pain intensity as described in inclusion criterion #2.
* Has painful diabetic sensorimotor polyneuropathy confirmed by modified Toronto Clinical Neuropathy Score (mTCNS) >5 at enrollment. The total score must include presence of foot pain (≥1) and sensory exam findings (≥ 2).
* Has hemoglobin A1c ≤10% as measured at enrollment.
* Is 22 years of age or older at the time of enrollment.
* Is an appropriate candidate for the surgical procedures required in this study based on the clinical judgment of the study physician.
* Is willing to and capable of giving written informed consent.
* Is willing and able to comply with study-related requirements and procedures and attend all scheduled visits.

Exclusion Criteria:

* Has a diagnosis of a lower limb mononeuropathy (e.g., causalgia, tibial or peroneal neuropathies), has had a lower limb amputation other than toes due to diabetes, or has large (≥3 cm) and/or gangrenous ulcers or active infection of the lower limbs.
* Has an average pain intensity of ≥ 3 out of 10 cm on the VAS in the upper limbs due to diabetic neuropathy at enrollment.
* Has a history of glycemia-related hospitalizations or emergency ward visits including ketoacidosis, hyperosmolar state, severe hypoglycemia in the previous 6 months.
* Uses anticoagulants or antiplatelet agents that cannot be temporarily discontinued prior to the procedure.
* Has unstable cardiovascular disease, including untreated cardiac arrhythmias, myocardial infarction within last 12 months, New York Heart Association (NYHA) Functional Class III or IV heart failure.
* Is currently prescribed a daily opioid dosage > 120 mg morphine equivalents.
* Has a medical condition or diagnosis that is inconsistent with the Senza System guidelines in the Physician's Manual or as per standard clinical practice.
* Has a medical condition or pain in other area(s), not intended to be treated in this study, that could interfere with study procedures, accurate pain reporting, and/or confound evaluation of study endpoints, as determined by the Investigator (such as primary headache, fibromyalgia, post-herpetic neuralgia, osteoarthritis, critical limb ischemia due to peripheral vascular disease or small vessel disease).
* Has prior experience with SCS, dorsal root ganglion (DRG) stimulation, peripheral nerve field stimulation (PNfS), or peripheral nerve stimulation (PNS) for chronic intractable pain.
* Has an existing drug pump and/or another active implantable device such as a pacemaker (ok to have an insulin pump or continuous glucose monitor that remains externalized).
* Has a condition currently requiring or likely to require the use of diathermy or MRI that is inconsistent with Senza System guidelines in the Physician's Manual.
* Has a life expectancy of less than one year.
* Has a local infection at the anticipated surgical entry site or an active systemic infection.
* Is pregnant or plans to become pregnant during the study (participants of child-bearing potential that are sexually active must use a reliable form of birth control).
* Has had within 6 months of enrollment a significant untreated addiction to dependency producing medications, alcohol or illicit drugs.
* Is concomitantly participating in another interventional clinical study.
* Is involved in an injury claim for study-related chronic pain that is under current litigation.
* Is a recipient of temporary Social Security Disability Insurance (SSDI) benefits due to study-related chronic pain.
* Has a pending or approved worker's compensation claim for study-related chronic pain.
* Has evidence of an active disruptive psychological or psychiatric disorder or other known condition significant enough to impact perception of pain, compliance with intervention and/or ability to evaluate treatment outcome, as determined by the investigator in the last 12 months.
* Has a BMI > 45 at enrollment.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2023-04-24 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Lower limb pain responder rate | 6 months
  The lower limb pain responder rate is the proportion of subjects who are pain responders, where a responder is defined as having at least 50% reduction in average lower limb pain score from baseline as measured on a 10-cm Visual Analog Scale (VAS, where a higher score indicates greater pain.

SECONDARY OUTCOMES:
Neurological improvement responder rate | 6 months
  The neurological improvement responder rate is the proportion of subjects who are neurological improvement responders, where a responder is defined as having a decrease of at least 3 points, excluding changes in foot pain under symptom scores, as assessed via the modified Toronto Clinical Neuropathy Score (mTCNS). The mTCNS assesses the severity of symptoms and sensory function loss associated with diabetic neuropathy. All symptom and sensory test scores are summed to provide a total mTCNS score for each assessment. The mTCNS has a maximum score of 33, where a higher score indicates greater neuropathy severity.
Lower limb pain responder rate at 3 months | 3 months
  The lower limb pain responder rate is the proportion of subjects who are pain responders, where a responder is defined as having at least 50% reduction in average lower limb pain score from baseline as measured on a 10-cm Visual Analog Scale (VAS), where a higher score indicates greater pain.
Percent change in lower limb pain intensity | 6 months
  Percent change in average lower limb pain intensity from baseline as measured on a 10-cm Visual Analog Scale (VAS), where a higher score indicates greater pain.
Percent change in PSQ-3 | 6 months
  Percent change in Pain and Sleep Questionnaire Three-Item Index (PSQ-3) score from baseline. PSQ-3 is a three-item questionnaire to assess the impact of chronic pain on sleep. Each question is answered on a 10-cm Visual Analog Scale (VAS), and the final score is the average of the three responses. A higher score indicates greater impact of chronic pain on sleep.
Average change in EQ-5D-5L index | 6 months
  Average change in EuroQol 5-dimension 5-level (EQ-5D-5L) index score from baseline. EQ-5D-5L measures the subject's health state as assessed in 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) each with 5 levels. The scores on these five dimensions can be presented as a health profile or can be converted to a single number summary called the "index value." A higher index score indicates higher quality of life.
Average change in NeuroQol | 6 months
  Average change in Neuropathy-Specific Quality of Life Questionnaire (NeuroQol) score from baseline. The NeuroQol measures a patient's perception of the impact diabetic peripheral neuropathy and foot ulcers on quality of life. Each question uses a 5-point Likert scale from 1 ("never") to 5 ("all the time") for frequency of symptoms. A higher NeuroQol value indicates greater impact of diabetic neuropathy on quality of life.
Average change in IENF density at the lower calf | 6 months
  Average change in intraepidermal nerve fiber (IENF) density at the lower calf from baseline. IENF is a measure of small nerve fiber density in the skin, with a higher value indicating greater density of nerve fibers.
Average change in mTCNS | 6 months
  Average change in the modified Toronto Clinical Neuropathy Score (mTCNS) from baseline. The mTCNS assesses the severity of symptoms and sensory function loss associated with diabetic neuropathy. All symptom and sensory test scores are summed to provide a total mTCNS score for each assessment. The mTCNS has a maximum score of 33, where a higher score indicates greater severity of neuropathy.
Average change in HbA1c | 6 months
  Average change in hemoglobin A1c (HbA1c) from baseline for patients with type 2 diabetes and HbA1c >= 8.0% at enrollment
Average change in body weight | 6 months
  Average change in body weight from baseline for patients with type 2 diabetes

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina
  - Touchstone Interventional Pain Center, Medford, Oregon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pop-Busui R, Petersen EA, Levy BL, Tesfaye S, Armstrong DG, Grunberger G, Boulton AJ, Bharara M, Edgar D, Azalde RP, Caraway D. Evaluating pain and neurological function with high frequency 10 kHz spinal cord stimulation in the treatment of painful diabetic neuropathy: design of a multicentre, randomised controlled trial (PDN-Sensory). BMJ Open. 2025 Nov 27;15(11):e101647. doi: 10.1136/bmjopen-2025-101647. PMID 41309477